CLINICAL TRIAL: NCT06170411
Title: A Multicenter, Double-blind, Parallel Design, Randomized, Placebo Controlled, Post-marketing Clinical Trial to Evaluate the Efficacy and Safety of Elexir (Trigeminal Nerve Electrical Stimulator) in Migraine Patients.
Brief Title: Post-marketing Clinical Trial of Elexir(Trigeminal Nerve Electrical Stimulator) for the Acute Treatment of Migraine
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Nu Eyne Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NE_MIG_002
Record Dates: First submitted 2023-11-08; First posted 2023-12-14 (Actual); Last update posted 2023-12-14 (Actual); Status verified 2023-11

CONDITIONS: Migraine
MeSH Terms: conditions — Migraine Disorders

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental Group (Experimental): 1-hour trigeminal nerve stimulation with the Elexir (program1), as acute treatment of an early stage migraine attack
  Interventions: Device: Elexir (program1)
- Control Group (Sham Comparator): 1-hour trigeminal nerve stimulation with the sham device, as acute treatment of an early stage migraine attack
  Interventions: Device: sham device

INTERVENTIONS:
Device: Elexir (program1) — The Elexir is an external cranial neurostimulator designed for supraorbital neurostimulation, also known as Trigeminal Nerve Stimulation. The Elexir will deliver trigeminal nerve stimulation.
  Arms: Experimental Group
Device: sham device — The sham device will deliver sham trigeminal nerve stimulation.
  Arms: Control Group

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of treating migraine in the acute phase by applying the acute mode (program 1) of Elexir (trigeminal nerve electrical stimulator) to patients with migraine.

DETAILED DESCRIPTION:
Written consent is obtained from the subjects before proceeding with this study. Afterwards, the selection/exclusion criteria are checked to determine whether they are suitable for participation in the study. Subjects who meet the final selection/exclusion criteria are randomly assigned and assigned to the test group or control group in a 1:1 ratio, clinical research coordinator will provide the subject with Investigational device to use at home and migraine diary, AE reporting form If migraine occurs within 8 weeks at home, the subject applies a investigational device (test device or control device) for 1 hour. A migraine diary is written after a migraine occurs and before starting a investigational device.

A migraine diary is written 1 and 2 hours after the start of application of the investigational device, and acute migraine treatment medications can be taken from that point on. Then, the subject writes migraine diary again 24 hours after starting to apply the investigational device.

Subjects who have applied the investigational device must visit the institution within 7 days after application and return the investigational device and the migraine headache.

If a subject does not occure a migraine within an 8-week period, subject must visit the institution and return the investigational device and migraine diary.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women19 to 65
2. A person who meet the ICHD-III (2018) criteria for migraine without aura and migraine with aura (ICHD-III sections 1.1, 1.2) However, typical aura, migraine with brainstem aura, and hemiplegic migraine without headache are excluded.
3. Having a history of migraine for more than 1 year
4. Migraine onset before the age of 50
5. Having between 2 and 8 migraine headaches* per month for 2 months in each of the two months prior to screening
6. A person who voluntarily agreed in writing to participate in this clinical trial

   * Migraine headache: Migraine attack lasting 4 to 72 hours (if untreated or inadequately treated), unilateral pulsating pattern, moderate or severe pain intensity (Grade 2 or 3 on the four-point Likert Scale), nausea, and /or headache accompanied by photophobia and phonophobia

Exclusion Criteria:

1. A person who has difficulty distinguishing between migraine and tension-type headache
2. A person who suffer from headaches more than 15 days a month
3. A person who underwents supraorbital nerve block within 4 months before the screening visit
4. A person who received Botox treatment within 4 months before the screening visit
5. Modification of a migraine prophylaxis treatment in the previous 3 months
6. A person diagnosed with other primary headaches excluding tension-type headaches less than 4 times a month
7. A person diagnosed with secondary headaches, including medication overuse headache
8. History of drug or alcohol abuse
9. A person judged to have other reasons for prohibiting the use of medical devices for clinical trials: A person implanted with metal or electronic devices such as head and neck implants, including deep brain stimulation devices, and persons implanted with implantable and wearable pacemakers. Those included in product precautions and contraindications (not applicable to dental implants)
10. Pregnant or lactating women
11. Among female subjects with childbearing potential, those who do not agree to maintain abstinence(not having sexual intercourse with the opposite sex) or to use contraception using a medically acceptable method* during the period of this clinical trial

    *Medically acceptable contraceptive methods: condoms, oral contraception for at least 3 months, use of injectable or insertable contraceptives, installation of an intrauterine contraceptive device, etc.
12. A person who participated in another clinical trial within 30 days of the screening visit
13. In other cases where the researcher determines that participation in the study is difficult (If you do not understand or cannot read the consent form for this clinical trial, etc.)

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-10-27 (Actual); Primary Completion 2024-08-01 (Estimated); Study Completion 2024-08-01 (Estimated)

PRIMARY OUTCOMES:
Changes in VAS score | 1 hour after beginning of the TNS session.
  Check the change in VAS socre 1 hour after beginning of the TNS session. The VAS scale consists of a total of 11 points, and the higher the score, the greater the pain.

SECONDARY OUTCOMES:
Pain Freedom | 1 hour, 2 hours after beginning of the TNS session.
  The percentage of patients having a reduction of a moderate or severe migraine headache (Grade 2 or 3) at baseline to no headache (Grade 0) at 1hour, 2 hours after beginning of the TNS session.
Most Bothersome Migraine-associated Symptom Freedom | 1 hour, 2 hours after beginning of the TNS session.
  The percentage of patients with absence, at 1 hour, 2 hours after the beginning of the TNS session, of the most bothersome migraine-associated symptom identified at baseline.
Pain Relief | 1 hour, 2 hours after beginning of the TNS session
  The percentage of patients having a reduction of a moderate or severe migraine headache (Grade 2 or 3) at baseline to a mild headache or to no headache (Grade 1 or 0) at 1 hour, 2 hours after beginning of the TNS session.
Percentage of Patients With Absence of Photophobia, Phonophobia, Nausea, Vomiting | 1 hour, 2 hours beginning of the TNS session
  The percentage of patients with absence of photophobia, phonophobia, nausea, vomiting at 1 hour, 2 hours after beginning of the TNS session.
Use of Rescue Medication Between 2 and 24 Hours | 2-24 hours after beginning of the TNS session
  The percentage of patients who took anti-migraine rescue medication between 2 and 24 hours after beginning of the TNS session.
Sustained Pain Freedom at 24 Hours | 24 hours after beginning of the TNS session
  The percentage of patients having no headache (Grade 0) at 2 hours, with no use of anti-migraine rescue medication and no relapse of headache pain within the 24 hours after the beginning of the TNS session.
Sustained Pain Relief at 24 Hours | 24 hours after beginning of the TNS session
  The percentage of patients having mild or no headache (Grade 1 or 0) at 2 hours, with no use of anti-migraine rescue medication and no relapse of headache pain within the 24 hours after the beginning of the TNS session.
Changes in headache intensity | 1 hour, 2 hours, 24 hours after beginning of the TNS session
  Check the change in Likert Scale 1 hour, 2 hours, 24 hours after beginning of the TNS session.
Rate of change in VAS score | 1 hour after beginning of the TNS session
  Check the rate of change in VAS socre 1 hour after beginning of the TNS session.

CONTACTS AND LOCATIONS:
Locations (2):
- South Korea (2):
  - Seoul National University Hospital, Seoul
  - Uijeongbu Eulji Medical Center, Eulji University, Uijeongbu-si

IPD SHARING:
Plan to Share IPD: No